CLINICAL TRIAL: NCT02703298
Title: A Phase I Safety and Pharmacokinetic Study of TRX-818 Administered Orally to Patients With Advanced Solid Tumors in Asians
Brief Title: Safety and Pharmacokinetic Study of TRX-818 in Asian Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVM-002
Record Dates: First submitted 2016-02-22; First posted 2016-03-09 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma; Advanced Cancer
Keywords: Advanced Solid Malignancy; Safety and Tolerability; Tumor Response; Oncology
MeSH Terms: conditions — Carcinoma; Neoplasms

ARMS (1):
- TRX-818 (Experimental)
  Interventions: Drug: TRX-818 capsules

INTERVENTIONS:
Drug: TRX-818 capsules

SUMMARY:
TRX-818 is a new small molecule chemical entity being developed as a potential anti-cancer therapeutic by TaiRx, Inc. TRX-818 is a potent anti-cancer agent in numerous human cancer cell lines. The objectives of this study are to determine the safety profile of TRX-818 including identification of dose limiting toxicity (DLT) and maximum tolerated dose (MTD) in Asians and determine the recommended dose and regimen(s) to initiate Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Tumor eligibility:

   Histologically or cytologically confirmed advanced, non resectable, and/or metastatic solid tumor refractory to standard of care therapy, or for whom no standard of care therapy is available, or who were not amenable to established forms of treatment.
2. Solid tumors must have measurable or evaluable disease as per Response Evaluation Criteria in Solid Tumors (RECIST v. 1.1). Target lesions that have been previously irradiated will not be considered measurable (lesion) unless increase in size is observed following completion of radiation therapy.
3. Female or male, 20 years of age or older.
4. ECOG performance status 0 to 2. Resolution of all acute toxic effects of prior therapy or surgical procedures to grade 1 (except alopecia).
5. Adequate organ function as defined by the following criteria: Serum aspartate transaminase (AST) and serum alanine transaminase (ALT) ≤3 x upper limit of normal (ULN), or AST and ALT ≤5 x ULN if liver function abnormalities are due to underlying malignancy; Total serum bilirubin ≤1.5 x ULN (except for patients with documented Gilbert's syndrome) ; Absolute neutrophil count (ANC) >= 1500/µL; Platelets >= 90,000/µL ; Hemoglobin >= 9.0 g/dL; Serum creatinine ≤2.0 x ULN
6. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
7. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with leukemia, lymphomas, multiple myeloma, or other type of hematologic cancers.
2. Major surgery, radiation therapy, or systemic anti-cancer therapy within 4 weeks of starting study treatment.
3. Prior high-dose chemotherapy requiring hematopoietic stem cell rescue.
4. Current treatment on another clinical trial.
5. Brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease unless appropriately treated and neurologically stable for at least 4 weeks.
6. Any of the following within the 12 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure, or cerebrovascular accident including transient ischemic attack; within 6 months prior to starting study treatment for pulmonary embolus. However, upon agreement between the investigator and sponsor, the 6 month post-event-free period for a patient with a pulmonary embolus can be waived if due to advanced cancer. Appropriate treatment with anticoagulants is permitted.
7. Hypertension that cannot be controlled by medications (>150/100 mmHg despite optimal medical therapy).
8. Current treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg PO daily for deep vein thrombosis prophylaxis is allowed).
9. Human immunodeficiency virus (HIV)-positive and is receiving anti-retroviral therapy.
10. Hepatitis B virus (HBV) or hepatitis C virus (HCV) with evidence of chronic active disease or receiving/requiring antiviral therapy.
11. History of receiving organ transplantation or immune disorders that require continuous immunosuppressant agent therapy.
12. Pregnancy or breastfeeding. Female patients must be surgically sterile or be postmenopausal, or must agree to the use of effective contraception during the period of therapy. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to enrollment. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
13. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that would impart, in the judgment of the investigator and/or sponsor, excess risk associated with study participation or study drug administration, which would make the patient inappropriate for entry into this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of TRX-818 in Asians | up to 28 days
  Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0.
Maximum tolerated dose (MTD) of TRX-818 in Asians | up to 28 days
  The MTD will be defined as the dose level at which at most one of six patients experiences a DLT after 28 days of treatment have occurred, with the next higher dose having at least 2/3 or 2/6 patients experiencing a DLT.

SECONDARY OUTCOMES:
Preliminary assessment of anti-tumor activity by Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) | up to 112 days
Composite measure of pharmacokinetics (PK) parameters of TRX-818: AUC(0-last) | Day 1, 8, 15 for Cycle 1 only(each cycle is 28 days)
  AUC(0-last): area under the plasma concentration versus time curve to the time of the last measurable concentration
Composite measure of pharmacokinetics (PK) parameters of TRX-818:Cmax | Day 1, 8, 15 for Cycle 1 only(each cycle is 28 days)
  Cmax: maximum plasma concentration
Composite measure of pharmacokinetics (PK) parameters of TRX-818: Tmax | Day 1, 8, 15 for Cycle 1 only(each cycle is 28 days)
  Tmax: time to maximum plasma concentration
Composite measure of pharmacokinetics (PK) parameters of TRX-818: T(1/2) | Day 1, 8, 15 for Cycle 1 only(each cycle is 28 days)
  T(1/2): terminal elimination half-life
Time to tumor progression (TTP) | up to 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Wu-Chou Su, M.D, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Tainan, Taiwan